CLINICAL TRIAL: NCT04613778
Title: Correction of Breech Presentation With Laser Acupuncture: a Randomized Controlled Trial
Brief Title: Correction of Breech Presentation With Laser Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000341A3
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Breech Presentation
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture (Experimental): Laser acupuncture with knee-chest position
  Interventions: Procedure: Laser acupuncture
- No intervention (No Intervention): usual care with knee-chest position

INTERVENTIONS:
Procedure: Laser acupuncture — Laser acupuncture is a low-level laser technique with no invasive procedure
  Arms: Laser acupuncture

SUMMARY:
Acupuncture-type interventions (such as moxibustion and acupuncture) at Bladder 67 (BL67, Zhiyin point) have been proposed to have positive effects on breech presentation. However, the role of laser acupuncture for Breech presentation remains unknown. The aim of this study is to evaluate the effectiveness and safety of laser acupuncture in correcting breech presentation.

ELIGIBILITY:
Inclusion Criteria:

* breech presentation or non-cephalic presentation
* gestation age 28~34 weeks
* singleton

Exclusion Criteria:

* uterus anomaly
* uterus tumors
* risk of preterm labor

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cephalic presentation at gestation age (GA) of 36 weeks | at gestation age (GA) 36 weeks
  numbers of cephalic presentation confirmed by ultrasound

SECONDARY OUTCOMES:
Cephalic presentation at labor | numbers of cephalic presentation at labor (an average of GA 38 weeks)
  confirmed by ultrasound

OTHER OUTCOMES:
adverse events | through study completion, an average of 6 weeks
preterm labor | through study completion, an average of 6 weeks
methods of delivery | at labor, an average of GA 38 weeks
  C/S or vaginal delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided